CLINICAL TRIAL: NCT01804075
Title: Evaluation of Efficacy of Methadone Versus Morphine for Treatment of Neonatal Abstinence Syndrome (NAS).
Brief Title: Comparison Between Methadone and Morphine for Neonatal Opiate Withdrawal
Acronym: NAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Maine Medical Center (Other)
Responsible Party: Principal Investigator, Mark S Brown, MD, Chief of Pediatric Service, Neonatalogy, Eastern Maine Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-1-M-185
Record Dates: First submitted 2012-11-06; First posted 2013-03-05 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-08

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: NAS; NICU; EMMC
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Methadone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- methadone (Active Comparator): Methadone (1 mg/mL) administered orally every 4 hours. The following is a dosing guide:
  NAS Score Methadone 8-12 0.05 mg/kg/dose >=13 0.1 mg/kg/dose
  1. Maximum dose of methadone will be 0.2 mg/kg/dose. (NeoFax)
  2. Additional doses, 0.05 mg/kg, may be given every 4 hours as needed and added to the next 24 hour's doses divided every 4 hours, until NAS scores are consistently <8 for 48 hours.
  3. If the maximum dose of methadone is reached and if withdrawal is not controlled, the infant will be started on clonazepam (0.005 mg/kg/dose q 12h) per current treatment.
  Interventions: Drug: Methadone
- morphine (Active Comparator): Morphine (1 mg/mL) administered orally every 4 hours. The following is a dosing guide:
  NAS Score Morphine 8-12 0.05 mg/kg/dose >=13 0.1 mg/kg/dose
  1. Maximum dose of morphine will be 0.2 mg/kg/dose. (NeoFax)
  2. Additional doses, 0.05 mg/kg, may be given every 4 hours as needed and added to the next 24 hour's doses divided every 6 hours, until NAS scores are consistently <8 for 48 hours.
  3. If the maximum dose of morphine is reached and if withdrawal is not controlled, the infant will be started on clonazepam (0.005 mg/kg/dose q 12h) per current treatment.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — To compare the duration of opiate medication treatment for babies on methadone versus those on morphine.
  Other Names: see arm/group descriptions
  Arms: methadone
Drug: Morphine — To compare the duration of opiate medication treatment for babies on methadone versus those on morphine.
  Other Names: see arm/group descriptions
  Arms: morphine

SUMMARY:
Hypothesis is that the effectiveness of opiate treatment with morphine will result in shorter duration of opiate medication treatment and fewer infants treated with a second drug.

DETAILED DESCRIPTION:
The purpose is to compare treatment of NAS with two different initial medications with primary outcome of (1) reducing the duration of opiate medication treatment and (2) reducing the number of infants treated with a second medication.

Design is a randomized, blinded comparison. The comparison is between methadone and morphine

Research Design:

a. Procedures: NAS scoring is currently done on infants meeting the inclusion criteria. NAS scores are done every 2 hours for 24 hours and then every 4 hours when awake after feeding for the duration of observation and treatment.

i. NAS scores may indicate more than withdrawal. Conditions such as colic (hypercaloric formula, transient lactose intolerance), reflux, diaper irritation, prenatal SSRI exposure, and nicotine withdrawal or baseline irritability may influence the variability of scores. Decisions based on the NAS scores should take into account these factors for the infant.

b. Emergence of symptom, dosing, and initiation of treatment: Withdrawal significant enough to warrant consideration for treatment is defined as 2 NAS scores >8. Once this threshold has been reached and consent obtained, the infant is randomized to treatment arm, stratified for prenatal exposure to methadone or buprenorphine. Twins will be randomized together to the same arm. The treatment arms are either: i. Methadone (1 mg/mL) or morphine (1 mg/mL) administered orally every 4 hours. The following is a dosing guide:

NAS Score Methadone or Morphine 8-12 0.05 mg/kg/dose >13 0.1 mg/kg/dose

1. Maximum dose of methadone or morphine will be 0.2 mg/kg/dose. (NeoFax)
2. Additional doses, 0.05 mg/kg, may be given every 12 hours as needed and added to the next 24 hour's doses divided every 4 hours, until NAS scores are consistently <8 for 48 hours.
3. If the maximum dose of methadone or morphine is reached and if withdrawal is not controlled, the infant will be started on clonazepam (0.005 mg/kg/dose q 12h) per current treatment.

   c. Tapering medications: When the infant has NAS scores consistently <8 for 36 hours: i.The taper will be on a daily basis of 10% of the final maintenance dose. Dosages will be decreased in a measured amount to maintain NAS scores <8. After the last dose, there will be a 24 to 36 hour observation period.

   d.Non-tolerance of tapering: Non-tolerance of tapering is defined as 2 NAS scores >8 during the 12 hour period prior to the next taper dose: i.The tapering should be stopped at the current level. ii.If necessary, an extra dose of methadone or morphine can be given and added to the next day's dose divided into 6 doses. If withdrawal re-emerges after this dose (2 NAS scores >8), then the maintenance dose should be increased back to the last level; an extra dose may be given up to 4 to 5 hours after the previous dose.

   iii. If an extra dose is not given, the wean schedule can be resumed after 24 hours of NAS scores <8; when dosing is resumed, the frequency should be changed to every 4 hours with the same total daily dose.

   e. Holding of doses: Methadone or morphine will be held for poor feeding, respiratory depression, or somnolence at any time in the protocol.

ELIGIBILITY:
Inclusion Criteria:

i. Evidence of opioid withdrawal clinically defined by at least 2 NAS scores > 8 in an 8 hour time period, AND

ii. Gestation => 35 weeks at entry defined by best obstetrical and physical exam criteria, AND

iii. Medically stable condition in the opinion of the attending neonatologist, other than opiate withdrawal, AND

iv. Mother on opiate replacement treatment therapy - methadone or buprenorphine.

Exclusion Criteria:

i. Gestation < 35 weeks at entry defined by best obstetrical and physical exam criteria.

ii. Hypoglycemia, hypomagnesaemia, or hypocalcemia until corrected,

iii. Serious medical illness such as sepsis, pneumonia, thyroid dysfunction, meningitis, intracranial hemorrhage, perinatal depression, or respiratory failure requiring admission to the NICU.

iv. Evidence of major congenital anomalies or genetic syndromes that impact the neonatal course

v. Mother consistently taking prescribed benzodiazepine at the time of delivery

Ages: 2 Hours to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Brown, MD, Principal Investigator — Eastern Maine Medical Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Methadone: Methadone (1 mg/mL) administered orally every 4 hours. The following is a dosing guide:
  NAS Score Methadone 8-12 0.05 mg/kg/dose >=13 0.1 mg/kg/dose
  1. Maximum dose of methadone will be 0.2 mg/kg/dose. (NeoFax)
  2. Additional doses, 0.05 mg/kg, may be given every 4 hours as needed and added to the next 24 hour's doses divided every 4 hours, until NAS scores are consistently <8 for 48 hours.
  3. If the maximum dose of methadone is reached and if withdrawal is not controlled, the infant will be started on clonazepam (0.005 mg/kg/dose q 12h) per current treatment.
  Methadone, Morphine: To compare the duration of opiate medication treatment for babies on methadone versus those on morphine.
- Morphine: Morphine (1 mg/mL) administered orally every 4 hours. The following is a dosing guide:
  NAS Score Morphine 8-12 0.05 mg/kg/dose >=13 0.1 mg/kg/dose
  1. Maximum dose of morphine will be 0.2 mg/kg/dose. (NeoFax)
  2. Additional doses, 0.05 mg/kg, may be given every 4 hours as needed and added to the next 24 hour's doses divided every 6 hours, until NAS scores are consistently <8 for 48 hours.
  3. If the maximum dose of morphine is reached and if withdrawal is not controlled, the infant will be started on clonazepam (0.005 mg/kg/dose q 12h) per current treatment.
  Methadone, Morphine: To compare the duration of opiate medication treatment for babies on methadone versus those on morphine.
Period: Overall Study
Arm/Group | Methadone | Morphine
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Morphine Treated: infants randomized to receive morphine as their primary treatment for withdrawal
- Methadone Treated: infants randomized to receive methadone as their primary treatment for withdrawal
- Total: Total of all reporting groups
Arm/Group | Morphine Treated | Methadone Treated | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: days] | 2.1 (1) | 2.3 (1.2) | 2.2 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Days of Treatment With Opioid Medication
Description: The length of time in days that the treatment opioid was used on a measured taper to ameliorate withdrawal signs
Time Frame: From date of randomization until the date of last opioid dose or date of death from any cause, whichever came first, assessed up to 12 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- Methadone-treated: group of infants randomized to receive methadone treatment for their withdrawal
- Morphine-treated: Group randomized to receive morphine treatment for their withdrawal
Arm/Group | Methadone-treated | Morphine-treated
Number analyzed (Participants) | 15 | 16
days | 13.9 (4.6) | 22.9 (9.7)

2. Secondary Outcome: Second Drug for Withdrawal
Description: Number of infants treated with a second drug to treat their withdrawal
Time Frame: From date of randomization until the date of last opioid dose or date of death from any cause or date of discharge, whichever came first, assessed up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone Treated | Morphine Treated
Number analyzed (Participants) | 15 | 16
Participants | 5 | 9
Statistical Analysis 1: Comparison: Methadone Treated vs Morphine Treated; Test type: Superiority; p = 0.6, Chi-squared

ADVERSE EVENTS:
Arm/Group | Methadone | Morphine
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No